CLINICAL TRIAL: NCT06726681
Title: Assessment of Intracranial Pressure Using Optic Nerve Sheath Diameter in Head Trauma in Assiut University Emergency Department
Brief Title: Assessment of Intracranial Pressure Using Optic Nerve Sheath Diameter in Head Trauma in Assiut University
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Abdelhameed sedeek khalid, Assessment of intracranial pressure using optic nerve sheath diameter in head trauma in Assiut University Emergency department, Assiut University
Other Study IDs: head trauma patient
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Head Trauma Injury
Keywords: optic nerve sheath diameter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- head trauma: Trauma patients admitted to Emergency department with a history of acute head injury and loss of consciousness

SUMMARY:
Clinical performance of optic nerve sheath diameter measurement using ultrasound in comparison of CT brain to measure the intra cranial pressure in head trauma

DETAILED DESCRIPTION:
Traumatic head injuries (THI) are one of the major causes of mortality and morbidity world wild. Head injuries contribute to almost 50% of all injuries. Nowadays, head injury has become one of the biggest issues of almost more than 57 million people in the whole world living with the neurological problem raised by TBI, in which 10 million people require hospital base care[1].

in many developing countries, head injury is one of the commonest life-threatening injuries among trauma victims[2]. In Egypt, injuries are many times larger than documented as a result of underreporting and misdiagnosis[3].

Elevated intracranial pressure (ICP) is a challenging and potentially fatal complication of acute head trauma. The elevation in intracranial pressure might lead to life-threatening conditions such as brainstem herniation and compromises cerebral perfusion. Early detection of raised intracranial pressure (RICP) is considered a better strategy to prevent secondary brain insults[2]. Early intervention in the form of either surgical evacuation of the space-occupying haematoma or medical management of the raised ICP is required, and cranial CT is necessary in deciding whether or not to operate. However, direct measurement of raised ICP requires an invasive procedure: the insertion of an ICP monitoring catheter. Some brain computed tomography (CT) findings, such as brain parenchymal swelling, midline shifting, and compressed basal cisterns, are traditionally used for the indirect measurement of raised ICP[4]. Although the invasive methods such as intraparenchymal and intra-ventricular devices are the reference standard for ICP monitoring but they not always used due to many causes such as unavailability of the technique expert in many hospitals, presence of contraindications (coagulopathy) and cost. In addition, they have serious complications such as intra-cranial hemorrhage, seizure and infection[5].

Some non-invasive methods for measuring ICP can be used as alternatives to invasive techniques, including transcranial Doppler, tympanic membrane displacement, optic nerve sheath diameter (ONSD), computed tomography (CT), magnetic resonance imaging (MRI), and fundoscopy [6]. These non-invasive techniques do not carry the risk of complications as with invasive methods. Recently, adult studies have reported that measuring ONSD with non-invasive imaging technologies such as CT, MRI and ultrasound can be used as an alternative method to evaluate increased ICP[7]. However, CT and MRI for ONSD measurements are time-consuming, costly and usually require patient transportation. Thus, ultrasound assessments of ONSD could be a better option because of the low cost and rapid bedside operation without the need for radiation exposure, especially for cases that are unstable and require real-time monitoring of ICP in an intensive care unit [8].

Several neuroimaging efforts have targeted novel methods for triaging head injury and early prognostication. The most popular, which is the ONSD measurement, has become a valuable adjunct to other clinical and laboratory prognostic indices, such as the Glasgow Coma Score (GCS)[9]. The measurement of ONSD can be performed as an alternative to invasive methods, because it can be performed bedside, with comparable results to invasive methods as well as a sensitivity and specificity of more than 90% [10].

The optic nerve sheath enclosing the optic nerve surrounds the optic subarachnoid space and is directly linked to the intracranial subarachnoid space. A rise in ICP pushes cerebrospinal fluid (CSF) from the intracranial cavity into the optic subarachnoid space with a resultant distension of the optic nerve sheath and its diameter. This uninterrupted connection provides easy access to measure ICP transmitted through the optic nerve sheath. ONSD assessment via ultrasonography is reflective of the variation in intracranial tension. The ONSD is known to increase within seconds of raised ICP, and this rise in ONSD is followed by a concurrent optic disk edema [11].

ONSD measurement can be performed using three methods: ultrasonography (USG), computed tomography (CT), and magnetic resonance imaging (MRI). In a meta-analysis that compared the usefulness of these three methods for ONSD measurement in cases of increased intracranial pressure, USG showed higher diagnostic accuracy than the other two methods [12]. In addition, because USG does not cause ionizing radiation exposure and can be easily performed at bedside in a short time and can be repeated, it is considered more advantageous than the other methods and is preferred more often in diagnostic studies[13].

This study is to determine the accuracy of optic nerve sheath dilatation, as measured by bedside ultrasonography, in predicting elevated ICP and the need for surgical intervention among people with head injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from > 18 years old. Both male and female patients. GCS<15 post injury or pt sent to CT scan by neurosurgery for Intracranial injury's Patients with no past or current neurological or neuro-ophthalmological diseases and normal neurological exams .

Exclusion Criteria:

* Pregnant women. Patients with severe orbital trauma. penetrating eye injury, or other ocular pathologies such as glaucoma, optic neuritis, central retinal vein/artery occlusion, retrobulbar hematoma or orbital cellulitis.

Patient with preexisting neurological diseases. Blind patients. Patients with cardiac arrest . Patients who refused participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: head trauma patient
Sampling Method: Non-Probability Sample
Enrollment: 143 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Optic nerve sheath diameter | baseline
  Optic nerve sheath diameter measurement inmm using ultrasound immediately before CT

SECONDARY OUTCOMES:
Trauma severity score 2-GCS 3_outcome of patient | baseline

IPD SHARING:
Plan to Share IPD: Undecided